CLINICAL TRIAL: NCT00950183
Title: Motorized Continuous Cold Therapy Versus Standard Post-op Icing Protocol for Two Foot and Ankle Procedures: An Evaluation of Narcotic Consumption, Pain, Wound Healing, and Patient Satisfaction
Brief Title: Motorized Continuous Cold Therapy Versus Standard Post-op Icing Protocol for Two Foot and Ankle Procedures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment feasability
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Collaborators: DJO Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 020723E
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2014-10

CONDITIONS: Narcotic Consumption; Pain; Wound Healing; Patient Satisfaction
Keywords: cryotherapy; postoperative pain; Iceman; primary first metatarsal osteotomy (PMO); lateral ankle ligament reconstruction (LAR)
MeSH Terms: conditions — Pain; Patient Satisfaction; Pain, Postoperative | interventions — Ice

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Foot and Ankle Surgery (Other): Please note that the study was terminated prior to randomization of patients.
  Interventions: Device: Iceman® Cold Therapy unit (djOrtho); Other: Ice

INTERVENTIONS:
Device: Iceman® Cold Therapy unit (djOrtho) — postoperative cold therapy
Other: Ice — postoperative cold therapy

SUMMARY:
This study will compares differences in pain level, narcotic consumption, wound healing, patient satisfaction in patients randomized to the Iceman® cold pack therapy system (djOrtho, Inc) versus those who use ice. This will be assessed postoperatively following the foot and ankle procedures primary first metatarsal osteotomy (PMO) or lateral ankle ligament reconstruction (LAR).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to have either lateral ankle ligament reconstruction (LAR) surgery or primary first metatarsal osteotomy surgery
* Patients who agree to be compliant and to keep a patient diary daily for 2 weeks and to return to the clinic for a 2 week postoperative follow- up appointment

Exclusion Criteria:

* Patients with Diabetes Mellitus, peripheral vascular disease, Reynauds Syndrome, hypersensitivity to cold
* Patients allergic to hydrocodone or oxycodone
* Patients who are unwilling to complete the patient diary and/or follow their specific cold therapy instructions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Anderson, MD, Principal Investigator — OrthoCarolina, PA
Locations (1):
- OrthoCarolina, PA, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated before patients were randomized to the treatment arms. Thus, it is not possible to report the results for the individual treatment arms.
Period: Overall Study
Arm/Group | Foot and Ankle Surgery
Started | 36
Completed | 0
Not Completed | 36

BASELINE CHARACTERISTICS:
Groups:
- Foot and Ankle Surgery: Our target enrollment was 82 participants. We only enrolled 36 participants. The study was terminated due to low enrollment. As a result, patients were never randomized.
Arm/Group | Foot and Ankle Surgery
Number analyzed (Participants) | 36
Age, Continuous [Mean (Full Range); unit: Years] | 56 [25 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Pain Scores
Time Frame: postop day 1 up to postop day 14
Population: Data not analyzed due to study termination
Arm/Group | Foot and Ankle Surgery
Number analyzed (Participants) | 0

2. Secondary Outcome: Narcotic Pain Medication Usage
Time Frame: postop day 1 up to postop day 14
Population: Data not analyzed due to study termination.
Arm/Group | Foot and Ankle Surgery
Number analyzed (Participants) | 0

3. Secondary Outcome: Patient Satisfaction
Time Frame: first postoperative visit (between postop day 10 and 14)
Population: Data not analyzed due to study termination
Arm/Group | Foot and Ankle Surgery
Number analyzed (Participants) | 0

4. Secondary Outcome: Surgical Complications
Time Frame: Day of Surgery
Population: Data not analyzed due to study termination
Arm/Group | Foot and Ankle Surgery
Number analyzed (Participants) | 0

5. Secondary Outcome: Postoperative Complications
Time Frame: postop day 1 up to postop day 14
Population: Data not analyzed due to study termination
Arm/Group | Foot and Ankle Surgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: There were no adverse events at time of study termination
Arm/Group | Foot and Ankle Surgery
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

LIMITATIONS AND CAVEATS:
The study was stopped due to poor enrollment. No results are available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No